CLINICAL TRIAL: NCT00694694
Title: A Randomized Trial of Azithromycin + Artesunate v Artemether-lumefantrine in Uncomplicated Malaria in Tanzanian Children.
Brief Title: Azithromycin + Artesunate v Artemether-lumefantrine in Uncomplicated Malaria.
Acronym: CAZAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITCRVG50
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2009-03

CONDITIONS: Malaria
Keywords: Malaria; Africa; Child
MeSH Terms: conditions — Malaria | interventions — Azithromycin; Artesunate; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1AZ+AQ (Experimental): Azithromycin + artesunate
  Interventions: Drug: azithromycin + artesunate
- 2AL (Active Comparator): Artemether-lumefantrine
  Interventions: Drug: artemether-lumefantrine

INTERVENTIONS:
Drug: azithromycin + artesunate — Azithromycin 20mg/kg per day for three days (total 60 mg/kg) Artesunate 4mg/kg per day for 3 days
  Other Names: zithromax
  Arms: 1AZ+AQ
Drug: artemether-lumefantrine — Tablets are fixed-dose combinations and contain 20mg artemether and 120mg lumefantrine.
  For children 5-14.9kg 1 tab 2x a day for 3 days For children 15-24.9kg 2 tablets 2x a day for 3 days For children 25-35kg 3 tablets 2x a day for 3 days
  Other Names: coartem; riamet
  Arms: 2AL

SUMMARY:
This trial sets out to determine whether the combination of azithromycin and artesunate (AZ+AS) is as good as the current standard treatment for uncomplicated malaria in Tanzania, artemether-lumefantrine (AL). There are two reasons this is important

1. there are only a limited range of drug combinations which work against malaria in this area of Tanzania
2. azithromycin has antimalarial properties, but is also a broad-spectrum antibiotic, so if the combination is an effective antimalarial it might have a place where there are no diagnostic facilities as syndromic treatment for fever.

Artesunate and azithromycin have both been used alone or in combination with other drugs in children in Tanzania for many years, and are considered safe. There is trial evidence for the effectiveness of this combination in adults in Asia, as well as in-vitro (laboratory) evidence that it works against the malaria parasite.

The trial randomizes children with non-severe malaria to the new combination AZ+AS or the standard care arm AL. The primary outcome is the parasitological failure rate by day 28- meaning do malaria parasites get cleared, and stay cleared for at least 28 days. Secondary outcomes include safety.

DETAILED DESCRIPTION:
Trial drugs. Artemether-lumefantrine (AL) has been selected to be the drug used to treat uncomplicated malaria in Tanzania. There is extensive efficacy, effectiveness and safety data on this combination from Tanzania. Artesunate is a key component of most ACTs. It should not be used as monotherapy, but is highly effective as an antimalarial when used in combination with another drug with antimalarial properties. There are now many years of experience of artesunate combinations on Africa and it appears safe in children. Azithromycin is licensed for use in childhood infections and trachoma. It is well tolerated and appears very safe in children; for example it does not have the effects of occasional bone-marrow toxicity seen with chroramphenicol, or the skin reactions sometimes seen with sulpha-drugs. It is active against the majority of childhood bacterial infections. There is extensive safety data on azithromycin, including data on azithromycin safety and tolerability in African children. Azithromycin has been shown to have significant antimalarial activity in vitro. There is good in vitro data on artemisinin + azithromycin combinations against malaria including tests for interactions . As a prophylactic drug against malaria azithromycin is effective in both West and East Africa. Azithromycin-artesunate has been used as an antimalarial drug combination in Asia. There is experience from small trials of combinations of artemisinin drugs and azithromycin to treat P. falciparum in Southeast Asia which were less effective than artesunate-mefloquine and artemether-doxycycline but several factors, especially the low doses of azithromycin used in two of these studies and patterns of antibiotic use locally may well have contributed to this; the combination appears safe . This contrasts with the evidence in East Africa that azithromycin is an effective antimalarial when used for prophylaxis, and there are several reasons why it may well be more effective in East Africa than in SE Asia.

Objectives. The overall study objectives will therefore be to compare the efficacy of azithromycin-artesunate and artemether-lumefantrine in the treatment of non-severe falciparum malaria in children in an area of high antimalarial drug resistance.

Specific objectives are i) to compare the effects of the drugs on parasitological failure rates at 28 days in each arm, both unadjusted and adjusting for reinfection judged by genotyping ii) to compare the drugs for clinical failure rate at 28 days. iii) to compare the drugs for clinical and parasitological failure at day 42. iv) to compare the drug combinations for adverse events and side effects v) to undertake a cost-effectiveness analysis of the two drug combinations.

Study design.

A randomised controlled trial of azithromycin-artesunate and artemether-lumefantrine for the treatment of non-severe falciparum malaria in children between 6 months and 5 years old.

The trial will be conducted among children attending the MCH clinic in one of the hospitals in the Tanga region (Muheza Designated District Hospital) with symptoms compatible with malaria. Those with malaria parasites in their blood smear will be considered for inclusion.

The trial

1. A randomised, open-label trial will be carried out. The slide reader assessing the primary endpoint will be blind to treatment allocation, and analysis performed by intention-to-treat.
2. All study drug regimens will be oral. After educating the patient on the need to complete the course prescribed by the clinician, drugs will be administered as direct observed therapy (DOT) by a nurse of the study team for morning doses and the evening dose (AL only) will be taken at home.

Screening.

Patients with non-severe (WHO definition) slide proven malaria with >2000 parasites/microL will be recruited from the Maternal and Child Health (MCH) clinic of Teule Hospital following initial pilot studies to identify and solve logistic or other problems.

Project nurses will interview parents/guardians of all febrile children and of those with a recent (past 48 hours) history of fever to exclude other causes of fever. Those who are clearly seriously unwell (unconscious, fitting etc) will be triaged immediately to the emergency admissions team. Those with a fever or history of fever will be referred for rapid diagnostic testing (RDT) with blood taken by fingerprick. A slide will be taken at the same time, to be used by the study team or hospital team if appropriate. If RDTs are positive a study slide will be made, stained and read and they will be referred to the study physician; if RDTs are negative to the Teule hospital doctor. Duplicate thick and thin blood smears will be made from all probable malaria cases, Giemsa stained at pH 7.2, and examined microscopically. All patients seen by the study team will be re-assessed by the physician of the study team to exclude concomitant infection(s).

Regimen allocation

Random number generated by the computer will be allocated to the two study regimens in blocks of random size. Patients consenting to participate in the study will be registered numerically as they present. The registration (enrolment) number of each patient will determine the drug regimen to be given. Registration numbers will correspond to sealed opaque envelopes with treatment allocation. Opening an envelope will be deemed to be randomisation, and intention to treat analysis will proceed on that basis

Once randomised, the child will be treated with the study drug they are allocated unless they withdraw or are withdrawn from the study.

Follow-up

Patients would be observed on days 0,1,2,7,14,28 and 42. Finger-prick for malaria blood slide, haemacue and filter paper blood specimen for genotyping will be taken on days 0, 2, 7, 14, 28 and 42 or any day the child presents unwell, and venous blood drawn for a full blood count and liver enzymes on days 0 and 14.

Rescue medication

Quinine at a dose of 10-mg/kg body weight for 7 days will be the rescue medication, as per Tanzanian national guidelines.

1. If patients are found to have deteriorating clinical condition in the presence of asexual parasites from days 0-3 of treatment this will be deemed an early treatment failure; they will be admitted for parenteral treatment.
2. If patients develop severe or complicated malaria (WHO) at any other stage they will be admitted for parenteral treatment.
3. Patients who recrudesce with or without symptoms during the study period will be treated with oral quinine and visited every day by VHCs to support the guardian and detect any problems early. If there is any sign of deterioration or unexpected side effects they will be admitted. At day 7 post commencing rescue treatment all patients will have a blood film; if this is positive they will be admitted for directly observed therapy.
4. Patients who recrudesce after quinine treatment will be treated as inpatients according to local guidelines.

Recrudescence versus reinfection.

Blood for PCR will be collected from all patients at enrolment and on follow-up as outlined above. PCR analysis of parasite genes will be performed only in patients with re-appearance of parasitaemia in order to differentiate between re-infection and recrudescence.

Adverse events If a patient is unable to tolerate the trial medication the reason for discontinuation will be recorded in the Clinical Record Form as an "adverse event" and alternative rescue medication initiated.

Any significant clinical or laboratory abnormality as judged by the senior attending physician (PI) will be recorded as an adverse event.

Assessment of efficacy; primary outcome: day 28 slide clearance

The day of first treatment is day 0. The day 28 slide clearance rate is the primary end point of therapeutic efficacy for this trial. It is the proportion of treated patients with no asexual parasitaemia double-read by microscopists blind to treatment allocation, and who did not receive rescue medication within that period.

Assessment of efficacy; secondary endpoints. All analysis intention-to treat unless otherwise specified.

i) Day 14 slide clearance rate by slides double-read blind to treatment allocation ii) Clinical failure rate on or by day 28 iii) Clinical failure rate on or by day 14 iv) Parasitological and clinical failure at day 42 v) Day 28 recrudescence rate assessed by PCR vi) Day 14 and 42 recrudescence rate assessed by PCR vii) Day 28 hemoglobin level viii) Differences in side effects/AE between groups ix) A per-protocol analysis for all day 14 and day 28 outcomes

ELIGIBILITY:
Inclusion Criteria:

Children with symptoms suggestive of malaria and

1. P.falciparum of at least 2000 parasites per microL of blood
2. are able to take study drugs by the oral route
3. are able to attend stipulated days for follow up clinic and provide specimens
4. have a parent or guardian who can give informed written/verbal consent to participate in the study
5. aged 6-59 months.

Exclusion Criteria:

1. severe and complicated forms of malaria (WHO, 2000)
2. a mixed plasmodial infection
3. a concomitant disease masking assessment of the treatment response (cases in whom advanced HIV infection is suspected will lead to be referred for HIV counseling).
4. recent effective full dose antimalarial treatment (within 7 days), excluding chloroquine, SP and AQ which have >70% failure in this district, or combinations of these.
5. known hypersensitivity to any of the trial drugs.
6. live too far away for reliable follow-up

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Parasitological failure by day 28 | Within 28 days of treatment.

SECONDARY OUTCOMES:
Combined clinical and parasitological outcome by day 42 | 42 days after treatment
Adverse events other than parasitologial failure. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Whitty, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Teule Hospital, Muheza, Tanga, Tanzania

REFERENCES:
- [Derived] Sykes A, Hendriksen I, Mtove G, Mandea V, Mrema H, Rutta B, Mapunda E, Manjurano A, Amos B, Reyburn H, Whitty CJ. Azithromycin plus artesunate versus artemether-lumefantrine for treatment of uncomplicated malaria in Tanzanian children: a randomized, controlled trial. Clin Infect Dis. 2009 Oct 15;49(8):1195-201. doi: 10.1086/605635. PMID 19769536